CLINICAL TRIAL: NCT02166528
Title: The Study of Susceptibility Genes Localization for Female Pelvic Floor Dysfunction
Brief Title: The Study of Genes Localization for Female Pelvic Floor Dysfunction
Acronym: PFD POP UI
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Zhiqing, Liang (Other)
Collaborators: Shenzhen Huada Genomics Co., Ltd. (Unknown)
Responsible Party: Sponsor-Investigator, Zhiqing, Liang, Director of Obstetrics and Gynecology, Third Military Medical University
Organization: Third Military Medical University (Other)
Other Study IDs: 002
Record Dates: First submitted 2014-02-10; First posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Female Pelvic Floor Dysfunction
Keywords: female pelvic floor dysfunction; pelvic organ prolaps; urinary incontinence; massively parallel sequencing
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The sample of blood, urine, cervical exfoliated cells and tissue of patients with POP, UI or genital tract injury should be used only in this research with informed consent. The remaining part will be Safekeeping. All information is strictly confidential.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- experiment group: patients with FPFD
- control group: patients without FPFD

SUMMARY:
Female pelvic floor dysfunction (FPD) is due to defects in the pelvic support structures, degradation, damage or dysfunction. The main problem of which is pelvic organ prolapse(POP), urinary incontinence(UI) and genital tract injury. Although it does not pose a serious threat to life, but affect the patient's quality of life seriously in the physical, psychological, social behavior and other aspects. With the growing aging population, the incidence rate has gradually increased, and increasing demands for people's quality of life simultaneously, more and more attention was raised to PFD as common chronic diseases.

In recent years, the basic research, epidemiology, prevention, diagnosis and treatment of PFD have made great progress, especially in developing gynecological urology theory and reconstructive pelvic surgery. But overall the basic research of PFD is lagging behind, especially susceptibility gene localization and functional studies did not get enough attention.

ELIGIBILITY:
Inclusion Criteria:

1. female aging from 30 to 70-year old;
2. preoperative diagnosis of gynecologic malignancies;
3. have the ability to comply with Research programs;
4. voluntarily participate in the study and signed an informed consent form

Exclusion Criteria:

1. patients with severe cardiovascular diseases, kidney, liver and other vital organs diseases, bone marrow disease and mental illness;
2. patients suffering from autoimmune diseases;
3. patients with acute infectious disease or infection early phase of infection;
4. patients with urinary tract infection;
5. patients with infection or erosion of ano-genital skin;
6. for any other reason, the researchers considered unsuitable for inclusion.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The experiment group are patients with PFD. While the control group are volunteer patients without PFD on the basis of informed consent.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
susceptibility genes localization | 4 years
  Based on high-throughput sequencing platform, we expect to screen out susceptibility genes location in PFD, providing theoretical basis for individualized prevention, intervention and treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynaecology, Southwest Hospital, Third Military, Chongqing, Chongqing Municipality, China